CLINICAL TRIAL: NCT04959604
Title: Lymph Node Mapping Via the Flourescent Dye ICG in Colon Cancer Through Preoperative Application
Brief Title: Lymph Node Mapping Via Flourescent Dye in Colon Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCLNM
Record Dates: First submitted 2021-06-30; First posted 2021-07-13 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Colon Carcinoma; Lymph Node Metastases
Keywords: indocyanine green; lymphatic mapping; fluorescence
MeSH Terms: conditions — Colonic Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Intervention Model Description: Intervention group. Participants will receive a state of the art surgical procedure with additional lymph node mapping
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICG-marked Colon Carcinoma (Experimental): The participants will receive an endoscopic marking via ICG preoperatively
  Interventions: Procedure: ICG-marking endoscopically

INTERVENTIONS:
Procedure: ICG-marking endoscopically — Preoperatively the participants will receive an endoscopic marking at four points around the tumour with the fluorescent dye indocyanine green.

SUMMARY:
The aim of the study is to evaluate whether lymph nodes draining the region of the carcinoma are located only inside the lines of standard resection or in some percentages are located outside as well. The visualized nodes draining the region of the carcinoma will be correlated to location, fluorescent yes/no and nodal positive/negative.

The draining lymph nodes will be visualized using the fluorescent dye indocyanine green.

The aim of the study is to evaluate whether lymph nodes draining the region of the carcinoma are located only inside the lines of standard resection or in some percentages are located outside as well. The visualized nodes draining the region of the carcinoma will be correlated to location, fluorescent yes/no and nodal positive/negative.

The draining lymph nodes will be visualized using the fluorescent dye indocyanine green.

DETAILED DESCRIPTION:
Participants with a diagnosed (andeno)carcinoma of the ascending, transverse, descending and sigmoid colon will be included. Preoperatively the participants will receive an indocyanine green(ICG) injection at four points around the tumour endoscopically. The ICG marking will take place one to five days prior to surgery. In the draining lymph nodes of the specific region the ICG will accumulate and thus visible via fluorescence-camera during the surgery.

Intraoperatively, the precise locations of all fluorescent nodes will be documented photographically. A standard resection and lymph node dissection will be conducted, potential fluorescent nodes outside the standard resection lines will additionally be resected. The fresh specimen will then be measured, the fluorescent nodes marked and after the pathologic examination the nodes will be correlated to location, fluorescent yes/no and nodal positive/negative.

The aim ist not the visualization of the Sentinel node or the directly draining lymphatic vessel but all the nodes draining the peritumorous region at the point of surgery.

ELIGIBILITY:
Inclusion Criteria:

* histologically diagnosed carcinoma of the ascending, transverse, descending or sigmoid colon.

Exclusion Criteria:

* not wanting to participate
* other carcinoma then adenocarcinoma
* endoscopic marking not possible

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Intraoperative ICG-positive lymph nodes in vivo after endoscopic marking of the tumour | intraoperative assessment
  Counting ICG-positive sites intraoperatively
Video-analysis of ICG-positive lymph nodes in vivo after endoscopic marking of the tumour | video-analysis within one week after surgery
  Counting ICG-positive sites video-analysis
Number of ICG-positive lymph nodes after endoscopic marking of the tumour | within one week after surgery
  Picking ICG-positive lymph nodes ex vivo in unfixed specimen, sending ICG positive nodes separately to pathological examination
Correlation of nodal-positive lymph nodes inside/outside the standard resection area | within one week after surgery
  ICG-positive sites outside standard resection area will be "cherry picked", sent to pathological examination separatively.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Perez, Prof. Dr., Principal Investigator — Dept of General Visceral and Thoracic Surgery
Locations (1):
- University of Hamburg Medical Institutions, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No
Available on reasonable request